CLINICAL TRIAL: NCT03546972
Title: Choosing Health and Cancer Risk Reduction Through Good Eating and Exercise
Brief Title: Diabetes Prevention Program With or Without Hunger Training in Helping to Lower Breast Cancer Risk in Obese Participants
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-0507; NCI-2018-01275 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0507 (Other: M D Anderson Cancer Center); R21CA215415 (NIH)
Record Dates: First submitted 2018-05-14; First posted 2018-06-06 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Deleterious BRCA1 Gene Mutation; Deleterious BRCA2 Gene Mutation; Ductal Breast Carcinoma In Situ; Obesity; Overweight; Premalignant Lesion
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (DPP) (Active Comparator): Participants take part in DPP once a week over 1 hour for 16 weeks.
  Interventions: Other: Behavioral, Psychological or Informational Intervention; Other: Questionnaire Administration
- Group B (DPP-HT) (Experimental): Participants take part in DPP once a week over 1 hour for 16 weeks and hunger training once a week during weeks 2-6.
  Interventions: Other: Behavioral, Psychological or Informational Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Other: Behavioral, Psychological or Informational Intervention — Take part in DDP
Other: Behavioral, Psychological or Informational Intervention — Take part in HT
  Arms: Group B (DPP-HT)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This pilot trial studies how well a diabetes prevention program with or without hunger training works in helping to lower breast cancer risk in obese participants. A diabetes prevention program involves learning about and receiving materials on different strategies to encourage weight loss, and hunger training involves learning how to recognize hunger. It is not yet known whether adding hunger training to a diabetes prevention program helps participants control their weight that could reduce the risk of some cancers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the feasibility of adding hunger training to the Diabetes Prevention Program (DPP) using the following criteria: accrual rates > 50%, attrition rates < 20% and, in the DPP-plus-hunger training (HT) group, training protocol adherence rates > 75%.

SECONDARY OBJECTIVES:

I. Estimate the magnitude of effect sizes and variation in outcome variables for the DPP-only and DPP-plus-HT interventions on changes in weight; in metabolic and breast cancer risk biomarkers (e.g., fasting insulin and blood glucose [BG] levels, levels of glycosylated hemoglobin, insulin resistance, adiponectin, interleukin-6, and C-reactive protein); and in proposed behavioral mediators (e.g., reduction in total energy intake, overall eating frequency, percent of eating events occurring at or below the average fasting blood BG level).

II. Examine the mediation effects of proposed mechanisms of the interventions related to individual-level behavioral measures of eating self-regulation on the proposed outcomes using a multimodal approach of validated questionnaires and reliable ecological momentary assessment method.

OUTLINE: Participants are randomized to 1 of 2 groups.

GROUP A: Participants take part in DPP once a week over 1 hour for 16 weeks.

GROUP B: Participants take part in DPP once a week over 1 hour for 16 weeks and hunger training once a week during weeks 2-6.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) >= 27 kg/m^2.
* At high risk of developing breast cancer defined by one or more of the following: Gail model lifetime risk > 20% or a 5 year risk >1.66%, a history of deleterious BRCA1/2 mutation or mantle radiation, a history of ductal cancer in situ, or a history of high risk premalignant breast lesion.
* 12 months without a period/menstrual cycle or having had a bilateral oophorectomy.
* Ability to take digital time stamped photos.
* Internet access (daily).
* Reports being proficient in English (can read/write and speak fluently).

Exclusion Criteria:

* Previous participation in this trial. Participation is defined as screening. Re-screening is not allowed except for individuals excluded for BMI. Patients previous screened as ineligible due to BMI are allowed to be re-screened and enrolled if eligible.
* Has a current measured BMI less than 27 kg/m^2.
* Reports being unwilling to use Continuous Glucose Monitor (CGM), which requires daily blood sampling by finger pricks.
* Currently being actively treated for cancer other than nonmelanoma skin cancer.
* Known inability to participate in the ongoing appointments for the four months of the study and scheduled follow-up tests.
* Reported current diagnosis or history of type I diabetes or type 2 diabetes.
* Reported use of oral antidiabetic agents (OADs).
* Current use of any drug (except metformin) or anticipated change in concomitant medication, which the investigator's opinion could interfere with the glucose metabolism (e.g. systemic corticosteroids).
* Previous or current treatment with any insulin regimen other than basal insulin, e.g. prandial or pre-mixed insulin (short term treatment due to intercurrent illness including gestational is allowed at the discretion for the investigator).
* Previous or current treatment with GLP-1 receptor agonists (e.g. exenatide, liraglutide).
* Fasting blood glucose level > 126 and glycosylated hemoglobin (HbA1c) > 7%.
* Subjects considered by the investigator as unsuitable for the study for reasons not otherwise stated.

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-12-17 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of adding hunger training (HT) to Diabetes Prevention Program (DPP) as assessed by recruitment rate | Up to 2 years
  Measured by percentage of participants who enroll in the study.
Feasibility of adding hunger training (HT) to Diabetes Prevention Program (DPP) as assessed by drop-out rates | Up to 2 years
  Measured by percentage of participants who leave the study.
Feasibility of adding hunger training (HT) to Diabetes Prevention Program (DPP) as assessed by completion rates | Up to 2 years
  Measured by percentage of participants who complete the study.

SECONDARY OUTCOMES:
Changes in weight loss | Baseline to 2 years
  Will use linear regression to study the effects of participant characteristics (i.e., weight history) and their interactions with the treatment groups.
Changes in metabolic and breast cancer risk biomarkers | Baseline to 2 years
  Biomarkers will be assessed through blood draws.
Changes in proposed behavioral mediators through survey | At baseline and at 16 weeks
  Eating patterns will be assessed through survey ASA24 (Automated Self-assessment).

CONTACTS AND LOCATIONS:
Overall Officials: Karen M Basen-Engquist, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Jospe MR, Liao Y, Giles ED, Hudson BI, Slingerland JM, Schembre SM. A low-glucose eating pattern is associated with improvements in glycemic variability among women at risk for postmenopausal breast cancer: an exploratory analysis. Front Nutr. 2024 Apr 10;11:1301427. doi: 10.3389/fnut.2024.1301427. eCollection 2024. PMID 38660060
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org